CLINICAL TRIAL: NCT00067418
Title: Spectroscopic Determination of Brain Tumor Cells
Brief Title: Light Scattering Spectroscopy to Determine Brain Tumors
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030270; 03-N-0270
Record Dates: First submitted 2003-08-18; First posted 2003-08-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Epilepsy, Temporal Lobe; Temporal Lobe
Keywords: Glioma; Brain Tumor; Spectroscopy
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Glioma; Brain Neoplasms

SUMMARY:
This study will use light scattering spectroscopy (LSS) to analyze brain tissue removed from patients during brain surgery to determine if this new technology can be used to differentiate between normal and cancerous cells. LSS focuses light on cells or tissues, and the way that light is reflected back from the tissues provides information about the size of cells and the density of the cell nuclei (the part of the cell that contains the genes).

Patients between 18 and 75 years of age with a known or suspected brain tumor and patients with temporal lobe epilepsy that does not respond to medication may be eligible for this study. (Examination of tissue from patients with epilepsy will allow comparison of tumor and non-tumor brain cells.) All patients must require surgery to treat their condition.

Participants will be admitted to the Clinical Center for 3 to 10 days for physical and neurological examinations, blood and urine tests, and other tests needed to prepare for surgery. They will then undergo surgery. A small amount of tissue removed during surgery for pathological review will be collected for use in this study.

Half of the tissue will be examined using LSS to help determine the size of the cell and its nucleus. Studies will be done to measure how many of the cells are actively dividing and which proteins are expressed more often in tumor cells compared with normal cells. This information may shed light on how tumor cells are different from normal cells.

Participants may be contacted for up to 3 years to follow their health status.

DETAILED DESCRIPTION:
Optical spectroscopy for detection of brain tumors and tumor margins has been shown to be of use in distinguishing gliomas and metastatic tumor cells from surrounding white matter. Optical spectroscopy has the potential to provide immediate and accurate diagnostic information about the nature and quantity of neoplastic cells, in a minimally-or non-invasive fashion. We propose to use a new method of optical spectroscopy, polarized light-scattering spectroscopy (LSS), which permits discrimination of malignant cancer cells from normal brain cells by virtue of alterations in the cytoplasmic and nuclear ratios of these cells.

Patients suspected of having, or with prior biopsy proof of, a WHO grade II-IV central nervous system (CNS) glial tumor(s); those with metastatic brain tumor; or patients with medically-refractory temporal lobe epilepsy with a presumed hippocampal source of seizures, who are seen in the Surgical Neurology Branch, NINDS, will be considered for entry into this study. Tissue samples of tumor or normal lateral temporal neocortex resected as part of standard care will be collected at surgery and utilized for research.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Radiographic evidence of primary glial neoplasm of the CNS (WHO grade II-IV) or any patient with a known primary neoplasm of the CNS; patients with a known or with radiographic evidence of resectable metastatic brain tumor(s); or patients with temporal lobe epilepsy (TLE) in whom resective surgery, which will include the lateral termporal neocortex, is indicated.
2. Informed consent from patients age 18 or older.
3. No racial or ethnic group or gender is excluded.
4. Pregnant women who require brain surgery may participate in this study.

EXCLUSION CRITERIA:

1. Inability to provide informed consent prior to surgery.
2. Medical conditions that cannot be corrected prior to surgery that would be standard contraindications for neurosurgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2003-08; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lacroix M, Abi-Said D, Fourney DR, Gokaslan ZL, Shi W, DeMonte F, Lang FF, McCutcheon IE, Hassenbusch SJ, Holland E, Hess K, Michael C, Miller D, Sawaya R. A multivariate analysis of 416 patients with glioblastoma multiforme: prognosis, extent of resection, and survival. J Neurosurg. 2001 Aug;95(2):190-8. doi: 10.3171/jns.2001.95.2.0190. PMID 11780887
- [Background] Louis DN, Pomeroy SL, Cairncross JG. Focus on central nervous system neoplasia. Cancer Cell. 2002 Mar;1(2):125-8. doi: 10.1016/s1535-6108(02)00040-5. No abstract available. PMID 12086870
- [Background] Silbergeld DL, Chicoine MR. Isolation and characterization of human malignant glioma cells from histologically normal brain. J Neurosurg. 1997 Mar;86(3):525-31. doi: 10.3171/jns.1997.86.3.0525. PMID 9046311